CLINICAL TRIAL: NCT02411435
Title: Phase I, Single-center, Open Label, Fixed-sequence Cross-over Study to Evaluate the Effect of Rifampin on the Pharmacokinetics of Oral Cabotegravir in Healthy Subjects
Brief Title: Effect of Rifampin (RIF) on the Pharmacokinetics (PK) of Oral Cabotegravir (CAB) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 117010
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: rifampin; drug interaction; pharmacokinetics; cabotegravir
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment A(CAB 30mg)+B (RIF 600mg)+C (CAB 30mg and RIF 600mg) (Experimental): Subjects will receive a single dose of CAB 30 mg on day 1. Subjects will then receive RIF 600 mg once daily on days 8-28 with co-administration of a single dose of CAB 30 mg on day 21.
  Interventions: Drug: CAB; Drug: RIF

INTERVENTIONS:
Drug: CAB — CAB 30 mg as 1 tablet will be administered orally with 240 mL of water in the fasted state.
Drug: RIF — RIF 600 mg as 2 capsules of 300 mg will be administered orally with 240 mL of water in the fasted state.

SUMMARY:
CAB is an integrase inhibitor that is currently in Phase 2 clinical trials for the treatment and prevention of human immunodeficiency virus-1 (HIV-1) infection. RIF, a rifamycin used for treatment of tuberculosis (common co-infection in HIV-infected subjects), is a known inducer of uridine diphosphate (UDP)-glucuronosyltransferases (UGTs) and Cytochrome P450 3A4 (CYP3A4). CAB is primarily metabolized via UGT1A1 and UGT1A9, thus a drug interaction between CAB and RIF is possible. This study will be a phase I, single-center, open label, fixed-sequence cross-over study to compare the single dose PK of CAB oral 30 milligrams (mg) when co-administered with RIF 600 mg once daily at steady-state to those of CAB oral 30 mg administered alone. Fifteen subjects are planned to be enrolled to obtain 12 evaluable subjects for this study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 18.5 - 31.0 kg/meter square (m^2) (inclusive).
* Male or female - A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: a) Non-reproductive potential defined as: Pre-menopausal females with one of the following [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy; b) Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause >40 milli-international units per mililiter (MIU/mL) and estradiol <40 picogram/milliliter (pg/mL) (<147 picomoles/liter [pmol/L]) is confirmatory]; c) Reproductive potential and agrees to follow one of the options listed in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until after the last dose of study medication and completion of the follow-up visit.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of clinically significant cardiovascular disease including: a) Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate <45 and >100 beats per minute for male subjects and <50 and >100 beats per minute for female subjects, QRS duration >120 millisecond (msec), and QT interval corrected by Fridericia's formula (QTcF) >450 msec; b) Evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes (except early repolarization); c) History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease; d) Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree (type II) or higher], Wolf Parkinson White [WPW] syndrome) which in the opinion of the principal Investigator and GSK Medical Monitor, will interfere with the safety for the individual subject; e) Sinus pauses >3 seconds; f) Any significant arrhythmia which, in the opinion of the principal Investigator and GSK Medical Monitor, will interfere with the safety for the individual subject; g) Non-sustained (>=3 consecutive ventricular ectopic beats) or sustained ventricular tachycardia.
* Subjects must abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* A history of regular use of tobacco, or nicotine-containing products within 30 days prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of Hepatitis B surface antigen (HBsAg), positive Hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. Hepatitis B core antibody (HBcAb) with negative hepatitis B surface antibody should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Plasma CAB maximum observed concentration after single dose administration (Cmax) | Days 1, 2, 3, 4, 6, 8, 21, 22, 23, 24, 26, and 28
  Plasma PK samples collected at the following time points: Period 1 pre-dose (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours post dose. Period 3 pre-dose Day 21 (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours (Day 8) post dose.
Plasma CAB area under the concentration versus time from time zero to infinity after single dose administration (AUC(0-∞)) | Days 1, 2, 3, 4, 6, 8, 21, 22, 23, 24, 26, and 28
  Plasma PK samples collected at the following time points: Period 1 pre-dose (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours post dose. Period 3 pre-dose Day 21 (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours (Day 8) post dose.

SECONDARY OUTCOMES:
Plasma CAB concentration at 24 hours post dose (C24) | Days 2 and 22
  Plasma PK samples collected at Period 1 24 hours post dose and at Period 3 24 hours post dose will be used to measure plasma CAB C24.
Plasma CAB AUC from time zero to last time point with measurable concentration after single dose administration (AUC (0-t)) | Days 1, 2, 3, 4, 6, 8, 21, 22, 23, 24, 26, and 28
  Plasma PK samples collected at the following time points: Period 1 pre-dose (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours post dose. Period 3 pre-dose Day 21 (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours (Day 8) post dose.
Plasma CAB time of occurrence of Cmax (tmax) and terminal phase half-life (t1/2) | Days 1, 2, 3, 4, 6, 8, 21, 22, 23, 24, 26, and 28
  Plasma PK samples collected at the following time points: Period 1 pre-dose (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours post dose. Period 3 pre-dose Day 21 (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours (Day 8) post dose.
Plasma CAB apparent clearance following oral dosing (CL/F) | Days 1, 2, 3, 4, 6, 8, 21, 22, 23, 24, 26, and 28
  Plasma PK samples collected at the following time points: Period 1 pre-dose (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours post dose. Period 3 pre-dose Day 21 (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 (Day 3), 72 (Day 4), 120 (Day 6), 168 hours (Day 8) post dose.
Number of subjects with adverse events (AEs) as a measure of safety and tolerability | Up to 42 days
  AEs will be collected from the start of study treatment until the follow-up contact
Concurrent medication as a measure of safety and tolerability | Up to 42 days
  Concurrent medication will be reviewed from the start of study treatment until the follow-up contact.
Clinical laboratory screens as a measure of safety and tolerability | Day -1, 8, 13, 20, 23, 25, 28, and follow-up (up to Day 42)
  Haematology, clinical chemistry, urinalysis and additional parameters will be tested.
Electrocardiogram (ECG) as a measure of safety and tolerability | Day 1, 20, 21, and 23
Vital signs assessments as a measure of safety and tolerability | Day 1, 8, 20, 21, 25, 26, 28, and follow-up (up to Day 42)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Ford SL, Sutton K, Lou Y, Zhang Z, Tenorio A, Trezza C, Patel P, Spreen W. Effect of Rifampin on the Single-Dose Pharmacokinetics of Oral Cabotegravir in Healthy Subjects. Antimicrob Agents Chemother. 2017 Sep 22;61(10):e00487-17. doi: 10.1128/AAC.00487-17. Print 2017 Oct. PMID 28739783